CLINICAL TRIAL: NCT05470881
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of PRO-201 Ophthalmic Solution Applied on the Ocular Surface of Healthy Volunteers.
Brief Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of Ophtalmic Solution PRO-201
Acronym: PRO-201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPH201-0521/I
Record Dates: First submitted 2022-03-23; First posted 2022-07-22 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, non-comparative, open, unicentric study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-201 (Experimental): A total of 29 anticipated healthy volunteers will be exposed to the investigation product.
  Interventions: Drug: Atropine Sulfate

INTERVENTIONS:
Drug: Atropine Sulfate — Administration of one drop QD on both eyes for 14 days.

SUMMARY:
Evaluation of the safety and tolerability of PRO-201 (0.01% sulfate atropine) after its instillation on the ocular surface of healthy volunteers through the following variables: unexpected adverse events incidence and photophobia (primary outcome variables); as well as pupillary diameter, expected adverse events incidence, best near corrected visual acuity (BNCVA), best corrected visual acuity (BCVA), intraocular pressure (IOP), corneal and conjunctival staining, heart rate, blood pressure and ocular confort index (OCI),

DETAILED DESCRIPTION:
A total of 29 healthy volunteers will be enrolled in this study. They will receive one drop of the investigation product PRO-201 (0.01% atropine sulfate) once a day (QD) for a total of 14 days on both eyes. A final safety call will be performed one week after the last day of product application.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically healthy
* Ability to voluntarily sign an informed consent form (ICF).
* Ability and willingness to comply with the scheduled visits according to the intervention plan and other procedures of the study.
* Age between 18 and 35.
* Absence of history of contact lens use.
* Women of childbearing age must agree to continue (starting ≥ 30 days previous to the ICF) the use of a hormonal contraception method of a intrauterine device (IUD) during the period of the study.
* Best corrected visual acuity (BVCA) of at least 20/30 (logMAR 0.2) or better in both eyes.
* Best near corrected visual acuity (BNVCA) of at least 20/25 (logMAR 0.1) or better in both eyes.
* Presenting vital signs within normal parameters.
* Presenting an IOP ≥10 and ≤ 21 mmHg

Exclusion Criteria:

* Using any kind of ophthalmic topical products.
* Presenting known allergy or intolerance to any ingrediente of atropine eyedrops or any other derivatives of antimuscarinic agents.
* Using any medication of herbolary products (plant extracts, infusions, naturist preparations, homeopathy, etc) through any route of administration
* For women: being pregnant, breastfeeding or planning to get pregnant during the period of the study.
* Having participated in any clinical study 90 days prior to the inclusion in this study.
* Having participated in this clinical study.
* Inability to follow the lifestyle considerations of this study.
* History of any chronic degenerative disease, including diabetes and hypertension.
* Presenting active inflammatory or infectious diseases when entering this study.
* Presenting unresolved lesions or trauma when entering this study.
* History of any ocular surgery.
* History of any surgery, non-ocular, within the previous 3 months of entering this studies.
* Being or having an direct family member (spouse, parent/legal guardian, sibling, etc) as employee of the investigation site or the sponsor, who participates directly in this study.

Elimination criteria:

* Withdraw of ICF.
* Adverse event, related or not to the investigation product, that according to the principal investigator and/or the sponsor may affect the integrity of the patient to continue safely with the study's procedures.
* Hypersensitivity or lack of tolerance to any of the ingredients used during the study's procedures (fluorescein, lissamine green, tetracaine, etc)
* Hypersensitivity or lack of tolerance to the investigation product.
* Presenting an adherence to treatment < 90%, as determined through the subjects diary.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IIMET Investigación e Innovación en Medicina Traslacional, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-201: A total of 29 anticipated healthy volunteers webe exposed to the investigation product (ITT population n=29) The PP population (subjects who finished the study without presenting any mayor deviations to protocol and adherence equal or higher to 90%) was comprised by 27 subjects. .
  Atropine Sulfate: Administration of one drop QD on both eyes for 14 days.
Period: Overall Study
Arm/Group | PRO-201
Started | 29
Completed | 27
Not Completed | 2
Not completed — Adherence under 90% | 2

BASELINE CHARACTERISTICS:
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.033 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 29
Intraocular pressure (IOP) [Mean (Standard Deviation); unit: mmhg] | 14.67 (2.67)

OUTCOME MEASURES:

1. Primary Outcome: Number of Unexpected Adverse Events
Description: The number of adverse events presented that are not previously described / known for the active substance in this pharmaceutic form and concentration.
Time Frame: Through Day 21 ± 1 (Safety Call)
Population: as for baseline characteristics
Measure: Number; unit: adverse events
Units Other Than Participants: Eyes
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
adverse events | 41

2. Primary Outcome: Number of Patients With Photophobia
Description: The number of cases of photophobia.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Participants
  Basal Visit: Photophobia | 0
  Basal Visit: No Photophobia | 29
  Visit 1: Photophobia | 5
  Visit 1: No Photophobia | 24
  Final visit: Photophobia | 2
  Final visit: No Photophobia | 27

3. Secondary Outcome: Pupillary Diameter
Description: Measurement of pupillary diameter after exposure to the investigation product.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: Only the right eyes of the participants were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Number analyzed (Eyes (right)) | 29
mm
  BV pupillary diameter | 3.44 (0.44)
  V1 pupillary diameter | 3.95 (0.60)
  FV pupillary diameter | 3.94 (0.52)

4. Secondary Outcome: Percentage of Expected Adverse Events
Description: The percentage of adverse events presented that are expected, or previously described / known for the active substance in this pharmaceutic form and concentration.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit), 21 ± 1 (Safety Call)
Measure: Number; unit: percentage
Units Other Than Participants: Eyes
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
percentage | 92.7

5. Secondary Outcome: Measurement of the Change in Best Near Corrected Visual Acuity (BCNVA)
Description: The change in BCNVA after exposure to investigation product, compared to basal value.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: Only the values obtained from the right eyes were analyzed for this variable.
Measure: Mean (Standard Deviation); unit: LogMAR (Snellen Chart)
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-201
Number analyzed (Participants) | 29
Number analyzed (Eyes (right)) | 29
LogMAR (Snellen Chart)
  BV BCNVA | 0.00 (0.02)
  V1 BCNVA | 0.00 (0.02)
  FV BCNVA | 0.01 (0.02)

6. Other Pre Specified Outcome: Changes in Intraocular Pressure (IOP)
Description: The change in IOP after exposure to investigation product, compared to basal value.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: Only the values obtained from the right eyes were analyzed for this variable. The evaluated population for this outcome measure was the PP population (subjects who finished the study without presenting any mayor deviations to protocol and adherence equal or higher to 90%).
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-201
Number analyzed (Participants) | 27
Number analyzed (Eyes (right)) | 27
mmHg
  VB IOP | 14.67 (2.67)
  V1 IOP | 14.04 (1.91)
  FV IOP | 14.02 (2.32)

7. Other Pre Specified Outcome: Number of Cases With Corneal and Conjunctival Staining With Fluorescein
Description: It was graded according to the Sjögren's International Clinical Collaboration Alliance (SICCA) Ocular Staining Score (CTO). According to the CTO, grade 0 corresponds to the absence of punctate epithelial erosions (PEE); grade 1 is defined as the presence of 1-5 EEPs; grade 2 corresponds to 6-30 EEP; and >30 EEP will be classified as grade 3. Additionally, one qualification point will be added if: 1) EEP is present in the central portion of the cornea with a diameter of 4mm; 2) filaments are observed and 3) confluent staining patches, including linear staining, are observed. A higher score is a worse outcome.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: as for outcome 6
Measure: Number; unit: Eyes (right)
Units Other Than Participants: Eyes (right)
Groups:
- PRO-201: A total of 29 anticipated healthy volunteers were be exposed to the investigation product (ITT population; n=29) Two reported adherence under 90% and were not included in the PP population (n=27)
  Atropine Sulfate: Administration of one drop QD on both eyes for 14 days.
Arm/Group | PRO-201
Number analyzed (Participants) | 27
Number analyzed (Eyes (right)) | 27
Eyes (right)
  BV corneal and conjunctival staining with fluorescein : Grade 0 | 27
  BV corneal and conjunctival staining with fluorescein : Grade 1 | 0
  V1 corneal and conjunctival staining with fluorescein : Grade 0 | 26
  V1 corneal and conjunctival staining with fluorescein : Grade 1 | 1
  FV corneal and conjunctival staining with fluorescein : Grade 0 | 26
  FV corneal and conjunctival staining with fluorescein : Grade 1 | 1

8. Other Pre Specified Outcome: Measurement of Vital Signs (Systolic Blood Pressure)
Description: The change in blood pressure after exposure to investigation product, compared to basal value.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: The evaluated population for this outcome measure was the PP population (subjects who finished the study without presenting any mayor deviations to protocol and adherence equal or higher to 90%).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-201
Number analyzed (Participants) | 27
mmHg
  BV Systolic Blood Pressure | 119.74 (8.73)
  V1 BV Systolic Blood Pressure | 120.96 (6.14)
  FV BV Systolic Blood Pressure | 119.41 (7.48)

9. Other Pre Specified Outcome: Measurement of Vital Signs (Heart Rate)
Description: The change in heart rate after exposure to investigation product, compared to basal value.
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pulse per minutes
Arm/Group | PRO-201
Number analyzed (Participants) | 27
pulse per minutes
  BV Heart Rate | 70.93 (6.62)
  V1 Heart Rate | 73.15 (9.51)
  FV Heart Rate | 74.93 (8.11)

10. Other Pre Specified Outcome: Value of the Ocular Comfort Index (OCI) Questionnaire.
Description: It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100). A higher score is a worse outcome.
  Similar to the index for ocular surface diseases, the ocular comfort index (OCI) evaluates symptoms. The ICO contains 6 items that focus on the discomfort associated with the ocular surface. Each of these questions has two parts, which inquire separately the frequency and severity of the symptoms. The evaluator will deliver the questionnaire to the subject and allow the subject to answer it calmly without any pressure and / or coercion, will only assist him if he has difficulty understanding any of the questions.
Time Frame: Days: 1 (Basal Visit), 16 ± 1 (Final Visit)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PRO-201
Number analyzed (Participants) | 27
scores on a scale
  BV OCI | 24.93 (9.46)
  FV OCI | 25.05 (10.39)

11. Other Pre Specified Outcome: Number of Cases With Corneal and Conjunctival Staining With Lissamine Green
Description: as for outcome 7
Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
Population: as for outcome 6
Measure: Number; unit: Eyes (right)
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-201
Number analyzed (Participants) | 27
Number analyzed (Eyes (right)) | 27
Eyes (right)
  BV Corneal and conjunctival staining with lissamine green : Grade 0 | 27
  BV Corneal and conjunctival staining with lissamine green : Grade 1 | 0
  BV Corneal and conjunctival staining with lissamine green : Grade 2 | 0
  V1 Corneal and conjunctival staining with lissamine green : Grade 0 | 23
  V1 Corneal and conjunctival staining with lissamine green : Grade 1 | 2
  V1 Corneal and conjunctival staining with lissamine green : Grade 2 | 2
  FV Corneal and conjunctival staining with lissamine green : Grade 0 | 26
  FV Corneal and conjunctival staining with lissamine green : Grade 1 | 1
  FV Corneal and conjunctival staining with lissamine green : Grade 2 | 0

ADVERSE EVENTS:
Time Frame: From day 1 (basal visit) to the safety call on day 21(±2 days)
Description: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Arm/Group | PRO-201
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 21/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO-201 (N=29)
Burning sensation (Eye disorders) | 9
Foreign body sensation (Eye disorders) | 2
irritation in the area of instillation (Eye disorders) | 10
Blurred vision (Eye disorders) | 7
Ocular hyperemia (Eye disorders) | 4
Pruritus (Eye disorders) | 3
Tearing (Eye disorders) | 3
Headache (Nervous system disorders) | 2
decreased visual acuity (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05470881/Prot_SAP_000.pdf